CLINICAL TRIAL: NCT02367885
Title: An Open-label, Multi-center, Phase 1/2 Study to Evaluate the Safety and Immunogenicity of an Intramuscular Injection of TAK-850 in Healthy Pediatric Subjects
Brief Title: Phase 1/2 Study of TAK-850 Intramuscular Injection in Healthy Pediatric Participants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TAK-850/CCT-101; U1111-1166-6015 (Registry Identifier: UTN (WHO)); JapicCTI-152807 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Results first posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-03

CONDITIONS: Influenza Infection
Keywords: Prevention
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAK-850 0.5 mL injection (13-19 years of age) (Experimental): Single intramuscular injection of TAK-850 0.5 mL in participants aged 13-19 years
  Interventions: Drug: TAK-850 0.5 mL injection
- TAK-850 0.5 mL injection (3-12 years of age) (Experimental): Two intramuscular injections of TAK-850 0.5 mL in participants aged 3-12 years old.
  Interventions: Drug: TAK-850 0.5 mL injection
- TAK-850 0.25 mL injection (6-35 months of age) (Experimental): Two intramuscular injections of TAK-850 0.25 mL in participants aged 6-35 months old.
  Interventions: Drug: TAK-850 0.25 mL injection

INTERVENTIONS:
Drug: TAK-850 0.5 mL injection — TAK-850 injection
  Arms: TAK-850 0.5 mL injection (13-19 years of age); TAK-850 0.5 mL injection (3-12 years of age)
Drug: TAK-850 0.25 mL injection — TAK-850 intramuscular injection
  Arms: TAK-850 0.25 mL injection (6-35 months of age)

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of an intramuscular injection of TAK-850 in healthy pediatric Japanese participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-850, that is under development as a vaccine for influenza infection. This study will evaluate the safety and immunogenicity of TAK-850 in healthy Japanese children when given as an intramuscular injection.

The study will enroll approximately 99 participants (33 per treatment group) to receive TAK-850 in open label fashion, The participants will be assigned to each treatment group as follows:

* a single intramuscular injection of TAK-850/0.5 mL in 13 to 19 years old healthy Japanese children,
* Two injections of TAK-850/0.5 mL in 3 to 12 years old healthy Japanese children,
* Two injections of TAK-850/0.25 mL in 6 to 35 months old healthy Japanese children.

The overall time to participate in this trial is 22 days (13-19 years old) or 43 days (6 months to 12 years old). Participants will make up to 2 visits (13-19 years old) or 3 visits (6 months to 12 years old) to the site.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator or the subinvestigator, the participant and/or his/her representative and his/her guardian is capable of understanding and complying with protocol requirements.
2. The participant's representative can sign and date a written, informed consent form prior to the initiation of any study procedures.
3. The participant is a healthy Japanese child.
4. The participant is aged 6 months to 19 years, inclusive, at the time of starting to receive the study vaccine.
5. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from signing of informed consent until 12 weeks after the administration.

Exclusion Criteria:

[Only for participants at the age of 6-35 months old]

1. The participant is a preterm newborn (gestational age was less than 37 weeks) or a low-birth-weight newborn (birth weight was less than 2500 g).
2. The participant has received any investigational compound within 4 months prior to the initial injection of study vaccine.
3. The participant has been vaccinated with seasonal influenza vaccine within 6 months prior to the initial injection of study vaccine.
4. The participant has a history of influenza infection within 6 months prior to the initial injection of study vaccine.
5. The participant is a study site employee, an immediate family member of such an employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling), or may consent under duress.
6. The participant has uncontrolled, clinically significant manifestations of neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, endocrine or other disorders, which may impact the ability of the participant to participate or potentially confound the study results.
7. The participant has an armpit temperature ≥ 37.5°C prior to the initial injection of study vaccine on Day 1.
8. The participant has any medically diagnosed or suspected immune deficient condition.
9. The participant has an immune compromising condition or disease, or is currently undergoing a form of treatment or was undergoing a form of treatment that can be expected to influence immune response within 30 days prior to the initial injection of study vaccine. Such treatments include, but are not limited to, systemic or high dose inhaled corticosteroids (> 800 μg/day of beclomethasone dipropionate or equivalent; the use of inhaled and nasal steroids that do not exceed this level will be permitted), radiation treatment or other immunosuppressive or cytotoxic drugs.
10. The participant has received antipyretics within 4 hours prior to the initial injection of study vaccine.
11. The participant has a history of Guillain-Barré Syndrome, demyelinating disorders (including acute disseminated encephalomyelitis [ADEM] and multiple sclerosis) or convulsions.
12. The participant has a functional or surgical asplenia.
13. The participant has a rash, other dermatologic conditions or tattoos which may interfere with the evaluation of injection site reaction as determined by the Investigator.
14. The participant has a history of, or is infected with the Hepatitis B Virus (HBsAgs), Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV).
15. The participant has a known hypersensitivity to any component of TAK-850.
16. The participant has a history of severe allergic reactions or anaphylaxis.
17. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the initial injection of study vaccine or is unwilling to agree to abstain from alcohol and drugs throughout the study.
18. The participant has received any blood products (e.g. blood transfusion or immunoglobulin) within 90 days prior to the initial injection of study vaccine.
19. The participant has received a live vaccine within 4 weeks (28 days) or an inactivated vaccine within 2 weeks (14 days) prior to the initial injection of study vaccine.
20. If female, the participant is pregnant or lactating or intending to become pregnant before signing informed consent, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
21. The participant has donated whole blood ≥ 200 mL within 4 weeks (28 days), ≥ 400 mL within 12 weeks (84 days), ≥ 800 mL within 52 weeks (364 days), or blood components within 2 weeks (14 days) prior to the initial injection of study vaccine.
22. In the opinion of the investigator or subinvestigator, the participant is unlikely to comply with protocol requirements or is considered ineligible for any other reason.

    -

Ages: 6 Months to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Takeda
Locations (2):
- Japan (2):
  - Chuou-ku, Tokyo
  - Setagaya-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in Japan from 14 February 2015 to 2 May 2015.
Pre-assignment Details: Healthy pediatric participants of age group 6 months-19 years were enrolled in 1 of the 3 treatment groups: TAK-850 0.25 milliliter (mL): 6 - 35 months; TAK-850 0.5 mL: 3-12 Years and TAK-850 0.5 mL: 13-19 Years.
Groups:
- TAK-850 0.25 mL: 6-35 Months: Participants aged 6 to 35 months received TAK-850 0.25 mL (15 microgram [mcg]/0.5 mL of hemagglutinin [HA] antigen per strain), injection, intramuscularly on Day 1 and 22 in a treatment period of 43 days.
- TAK-850 0.5 mL: 3-12 Years: Participants aged 3 to 12 years received TAK-850 0.5 mL (15 mcg/0.5 mL of HA antigen per strain), injection, intramuscularly on Day 1 and 22 in a treatment period of 43 days.
- TAK-850 0.5 mL: 13-19 Years: Participants aged 13 to 19 years received TAK-850 0.5 mL (15 mcg/0.5 mL of HA antigen per strain), injection, intramuscularly on Day 1 in a treatment period of 22 days.
Period: Overall Study
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Started | 33 | 33 | 33
Completed | 31 | 33 | 33
Not Completed | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study vaccination.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years | Total
Number analyzed (Participants) | 33 | 33 | 33 | 99
Age, Customized [Number; unit: participants]
  6-35 Months | 33 | 0 | 0 | 33
  3-12 Years | 0 | 33 | 0 | 33
  13-19 Years | 0 | 0 | 33 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 19 | 50
  Male | 18 | 17 | 14 | 49
Region of Enrollment [Number; unit: participants]
  Japan | 33 | 33 | 33 | 99
Hemagglutination Inhibition (HI) (Egg-derived) - A/H1N1 Titer at Day 1(Pre-vaccination) [Number; unit: participants] — Number of participants with values of HI antibody titer for A/H1N1 strain pre-vaccination at Day 1 were reported.
  participants
    Less Than (<) 40 Titer | 31 | 6 | 14 | 51
    Greater Than or Equal to (>=) 40 Titer | 2 | 27 | 19 | 48
Hemagglutination Inhibition (HI) (Egg-derived) - A/H3N2 Titer at Day 1 (Pre-vaccination) [Number; unit: participants] — Number of participants with values of HI antibody titer for A/H3N2 strain pre-vaccination at Day 1 were reported.
  participants
    <40 Titer | 26 | 16 | 15 | 57
    >=40 Titer | 7 | 17 | 18 | 42
Hemagglutination Inhibition (HI) (Egg-derived) - B Titer at Day 1 (Pre-vaccination) [Number; unit: participants] — Number of participants with values of HI antibody titer for B strain pre-vaccination at Day 1 were reported.
  participants
    <40 Titer | 33 | 33 | 26 | 92
    >=40 Titer | 0 | 0 | 7 | 7
Influenza Infection within 5 years [Number; unit: participants]
  Infection occurred | 2 | 16 | 7 | 25
  Infection did not occur | 31 | 17 | 26 | 74
Administration of Antipyretics [Number; unit: participants]
  Antipyretics administered | 2 | 1 | 1 | 4
  Antipyretics not administered | 31 | 32 | 32 | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Events (AEs) for 6-35 Months Old Group
Description: Local reactions and systemic events were recorded using a diary. Number of participants with local reactions (Injection site tenderness, Injection site ecchymosis, Irritability postvaccinal) and systemic events (Pyrexia, sweaty, vomiting, crying abnormal, inappetence, somnolence, sleeplessness) were reported. Participants may be represented in more than 1 category.
Time Frame: Up to 21 days after any vaccination
Population: Safety analysis set included all participants who received at least 1 dose of study vaccination.
Measure: Number; unit: participants
Arm/Group | TAK-850 0.25 mL: 6-35 Months
Number analyzed (Participants) | 33
participants
  Injection site tenderness | 3
  Injection site ecchymosis | 4
  Pyrexia | 12
  Sweaty | 2
  Vomiting | 6
  Irritability postvaccinal | 2
  Crying abnormal | 2
  Inappetence | 3
  Somnolence | 5
  Sleeplessness | 2

2. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Events (AEs) for 3-12 Years Old Group and 13-19 Years Old Group
Description: Local reactions and systemic events were recorded using a diary. Number of participants with local reactions (Injection site pain, Injection site redness, Injection site swelling, Injection site induration, Injection site tenderness, Injection site ecchymosis) and systemic events (Pyrexia, malaise, chills, fatigue, headache, sweaty, myalgia, nausea, vomiting) were reported. Participants may be represented in more than 1 category.
Time Frame: Up to 21 days after any vaccination
Population: Safety analysis set included all participants who received at least 1 dose of study vaccination.
Measure: Number; unit: participants
Arm/Group | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33 | 33
participants
  Injection site pain | 19 | 8
  Injection site redness | 6 | 1
  Injection site swelling | 6 | 3
  Injection site induration | 3 | 2
  Injection site tenderness | 23 | 18
  Injection site ecchymosis | 1 | 0
  Pyrexia | 3 | 1
  Malaise | 5 | 3
  Chills | 1 | 0
  Fatigue | 4 | 2
  Headache | 1 | 1
  Sweaty | 1 | 0
  Myalgia | 3 | 1
  Nausea | 0 | 1
  Vomiting | 2 | 0

3. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly; or a medically important event. AEs included both SAE and non-SAE.
Time Frame: Up to 21 days after any vaccination
Population: Safety analysis set included all participants who received at least 1 dose of study vaccination.
Measure: Number; unit: participants
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33 | 33 | 33
participants
  AEs | 24 | 29 | 24
  SAEs | 0 | 1 | 0

4. Primary Outcome: Percentage of Participants With Seroprotection in Hemagglutination Inhibition (HI) Antibody Titer (Egg-Derived Antigen) of >=40: 21 Days After the Vaccination for 13-19 Years Old Group
Description: Seroprotection rate was measured by HI antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination for the age group of 13-19 years. Seroprotection rate was defined as the percentage of participants with HI antibody titer of >=40.
Time Frame: Day 22 (21 days after Vaccination)
Population: All participants included in the full analysis set (FAS) (all participants who received at least 1 dose of study vaccination) who had data available for specified strain at specified post-baseline time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33
percentage of participants
  A/H1N1 Strain | 97.0 [84.241 to 99.923]
  A/H3N2 Strain | 93.9 [79.774 to 99.257]
  B Strain | 66.7 [48.173 to 82.039]

5. Primary Outcome: Percentage of Participants With Seroprotection in HI Antibody Titer (Egg-Derived Antigen) of >=40: 21 Days After the Second Vaccination for 6-35 Months Old Group and 3-12 Years Old Group
Description: Seroprotection rate was measured by HI antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after second vaccination for two age groups: 6-35 months and 3-12 years. Seroprotection rate was defined as the percentage of participants with HI antibody titer of >=40.
Time Frame: Day 43 (21 days after Vaccination 2)
Population: All participants included in the FAS (all participants who received at least 1 dose of study vaccination) who had data available for specified strain at specified post-baseline time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years
Number analyzed (Participants) | 33 | 33
percentage of participants
  A/H1N1 Strain (n=31, 31) | 87.1 [70.166 to 96.370] | 100 [88.781 to 100.000]
  A/H3N2 Strain (n=31, 31) | 71.0 [51.964 to 85.777] | 90.3 [74.246 to 97.958]
  B Strain (n=31, 31) | 9.7 [2.042 to 25.754] | 45.2 [27.316 to 63.966]

6. Primary Outcome: Percentage of Participants With Seroconversion in Hemagglutination Inhibition (HI) Antibody Titer (Egg-Derived Antigen): 21 Days After the Vaccination for 13-19 Years Old Group
Description: Seroconversion rate was measured by HI antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination for the age group of 13-19 years. Seroconversion rate was defined as the percentage of participants achieving a minimal 4-fold increase from baseline (with a baseline HI antibody titer of >=10), or achieving a HI antibody titer of >=40 (with a baseline HI antibody titer of <10) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain).
Time Frame: Day 22 (21 days after Vaccination)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33
percentage of participants
  A/H1N1 Strain | 66.7 [48.173 to 82.039]
  A/H3N2 Strain | 45.5 [28.107 to 63.649]
  B Strain | 45.5 [28.107 to 63.649]

7. Primary Outcome: Percentage of Participants With Seroconversion in HI Antibody Titer (Egg-Derived Antigen): 21 Days After the Second Vaccination for 6-35 Months Old Group and 3-12 Years Old Group
Description: Seroconversion rate was measured by HI antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after second vaccination for two age groups: 6-35 months and 3-12 years. Seroconversion rate was defined as the percentage of participants achieving a minimal 4-fold increase from baseline (with a baseline HI antibody titer of >=10), or achieving a HI antibody titer of >=40 (with a baseline HI antibody titer of <10) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain).
Time Frame: Day 43 (21 days after Vaccination 2)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years
Number analyzed (Participants) | 33 | 33
percentage of participants
  A/H1N1 Strain (n=31, 31) | 80.6 [62.527 to 92.548] | 71.0 [51.964 to 85.777]
  A/H3N2 Strain (n=31, 31) | 58.1 [39.076 to 75.452] | 54.8 [36.034 to 72.684]
  B Strain (n=31, 31) | 9.7 [2.042 to 25.754] | 45.2 [27.316 to 63.966]

8. Primary Outcome: Geometric Mean Fold Increase (GMFI) in HI Antibody Titer (Egg-Derived Antigen) From Baseline to 21 Days After the Vaccination for 13-19 Years Old Group
Description: GMFI from baseline in HI antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination for the age group of 13-19 years.
Time Frame: Day 22 (21 days after Vaccination)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33
fold increase
  A/H1N1 Strain | 13.53 [6.340 to 28.852]
  A/H3N2 Strain | 3.66 [2.212 to 6.050]
  B Strain | 3.68 [2.374 to 5.698]

9. Primary Outcome: GMFI in HI Antibody Titer (Egg-Derived Antigen) From Baseline to 21 Days After the Second Vaccination for 6-35 Months Old Group and 3-12 Years Old Group
Description: GMFI from baseline in HI antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after second vaccination for two age groups: 6-35 months and 3-12 years.
Time Frame: Day 43 (21 days after Vaccination 2)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years
Number analyzed (Participants) | 33 | 33
fold increase
  A/H1N1 Strain (n=31, 31) | 14.23 [8.856 to 22.857] | 6.15 [4.076 to 9.284]
  A/H3N2 Strain (n=31, 31) | 5.85 [3.728 to 9.183] | 4.73 [2.882 to 7.764]
  B Strain (n=31, 31) | 1.32 [0.958 to 1.825] | 2.86 [1.823 to 4.489]

10. Secondary Outcome: Percentage of Participants With Seroprotection in HI Antibody Titer (Egg-Derived Antigen) of >= 40: 21 Days After the First Vaccination for 6-35 Months Old Group and 3-12- Years Old Group
Description: Seroprotection rate was measured by HI antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after first vaccination for two age groups: 6-35 months and 3-12 years. Seroprotection rate was defined as the percentage of participants with HI antibody titer of >=40.
Time Frame: Day 22 (21 days after Vaccination 1)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years
Number analyzed (Participants) | 33 | 33
percentage of participants
  A/H1N1 Strain (n=32, 32) | 15.6 [5.275 to 32.788] | 93.8 [79.193 to 99.234]
  A/H3N2 Strain (n=32, 32) | 28.1 [13.746 to 46.747] | 75.0 [56.595 to 88.538]
  B Strain (n=32, 32) | 6.3 [0.766 to 20.807] | 46.9 [29.094 to 65.256]

11. Secondary Outcome: Percentage of Participants With Seroconversion in HI Antibody Titer (Egg-Derived Antigen): 21 Days After the First Vaccination for 6-35 Months Old Group and 3-12 Years Old Group
Description: Seroconversion rate was measured by HI antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after the first vaccination for two age groups: 6-35 months and 3-12 years. Seroconversion rate was defined as the percentage of participants achieving a minimal 4-fold increase from baseline (with a baseline HI antibody titer of >=10), or achieving a HI antibody titer of >=40 (with baseline HI antibody titer of <10) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain).
Time Frame: Day 22 (21 days after Vaccination 1)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years
Number analyzed (Participants) | 33 | 33
percentage of participants
  A/H1N1 Strain (n=32, 32) | 9.4 [1.977 to 25.023] | 53.1 [34.744 to 70.906]
  A/H3N2 Strain (n=32, 32) | 15.6 [5.275 to 32.788] | 37.5 [21.100 to 56.308]
  B Strain (n=32, 32) | 6.3 [0.766 to 20.807] | 46.9 [29.094 to 65.256]

12. Secondary Outcome: GMFI in HI Antibody Titer (Egg-Derived Antigen) From Baseline to 21 Days After the First Vaccination for 6-35 Months Old Group and 3-12 Years Old Group
Description: GMFI from baseline in HI antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after first vaccination for two age groups: 6-35 months and 3-12 years.
Time Frame: Day 22 (21 days after Vaccination 1)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years
Number analyzed (Participants) | 33 | 33
fold increase
  A/H1N1 Strain (n=32, 32) | 1.41 [1.059 to 1.888] | 5.36 [3.221 to 8.916]
  A/H3N2 Strain (n=32, 32) | 1.58 [1.158 to 2.145] | 3.15 [2.020 to 4.917]
  B Strain (n=32, 32) | 1.22 [0.907 to 1.628] | 3.22 [1.972 to 5.260]

13. Secondary Outcome: Geometric Mean Titer (GMT) of HI Antibody Titer (Egg-Derived Antigen)
Description: GMT of HI antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after each vaccination. Analysis after Vaccination 2 is only applicable for 6-35 Months old group and 3-12 Years old group.
Time Frame: Day 22 (21 days after Vaccination 1 for all groups), Day 43 (21 days after Vaccination 2 for 6-35 months old group and 3-12 years old group)
Population: All participants included in FAS (all participants who received at least 1 dose of study vaccination) who had available data for specified strain at specified post-baseline time points.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33 | 33 | 33
titer
  A/H1N1: 21 days after Vaccination 1 (n=32,32,33) | 8.78 [5.872 to 13.132] | 583.71 [351.985 to 967.995] | 558.32 [391.258 to 796.705]
  A/H1N1: 21 days after Vaccination 2 (n=31,31, 0) | 88.96 [57.072 to 138.677] | 773.95 [576.157 to 1039.645] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  A/H3N2: 21 days after Vaccination 1 (n=32,32,33) | 17.56 [9.046 to 34.086] | 87.24 [47.894 to 158.908] | 133.14 [86.409 to 205.133]
  A/H3N2: 21 days after Vaccination 2 (n=31,31, 0) | 66.90 [38.136 to 117.347] | 127.94 [76.820 to 213.092] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  B: 21 days after Vaccination 1 (n=32,32,33) | 6.08 [4.535 to 8.141] | 16.82 [10.192 to 27.751] | 28.58 [18.421 to 44.351]
  B: 21 days after Vaccination 2 (n=31,31,0) | 6.61 [4.790 to 9.127] | 14.96 [9.400 to 23.792] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.

14. Secondary Outcome: Percentage of Participants With Seroprotection in Single Radial Hemolysis (SRH) Antibody Titer (Egg- Derived Antigen) of >=25 Square Millimeter (mm^2)
Description: Seroprotection rate was measured by SRH antibody titer (egg- derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after each vaccination for all groups. Seroprotection rate was defined as the percentage of participants with SRH antibody titer of >=25 mm^2. Analysis after Vaccination 2 is only applicable for 6-35 months old group and 3-12 years old group.
Time Frame: as for outcome 13
Population: All participants included in the FAS (all participants who received at least 1 dose of study vaccination) who had data available for specified strain at specified post-baseline time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33 | 33 | 33
percentage of participants
  A/H1N1: 21 days after Vaccination 1 (n=32, 32, 33) | 9.4 [1.977 to 25.023] | 90.6 [74.977 to 98.023] | 100 [89.424 to 100.000]
  A/H1N1: 21 days after Vaccination 2 (n=29, 31, 0) | 79.3 [60.275 to 92.006] | 100 [88.781 to 100.000] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  A/H3N2: 21 days after Vaccination 1 (n=32, 32, 33) | 28.1 [13.746 to 46.747] | 78.1 [60.027 to 90.723] | 97.0 [84.241 to 99.923]
  A/H3N2: 21 days after Vaccination 2 (n=29, 31, 0) | 79.3 [60.275 to 92.006] | 93.5 [78.578 to 99.209] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  B: 21 days after Vaccination 1 (n=32, 32, 33) | 15.6 [5.275 to 32.788] | 78.1 [60.027 to 90.723] | 97.0 [84.241 to 99.923]
  B: 21 days after Vaccination 2 (n=29, 31, 0) | 48.3 [29.449 to 67.469] | 87.1 [70.166 to 96.370] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.

15. Secondary Outcome: Percentage of Participants With Seroconversion in SRH Antibody Titer (Egg-Derived Antigen)
Description: Seroconversion rate was measured by SRH antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after each vaccination for all groups. Seroconversion rate was defined as the percentage of participants achieving a minimal 50% increase from baseline (with a baseline SRH antibody titer of >4 mm^2) or achieving a SRH antibody titer of >=25 mm^2 (with baseline SRH antibody titer of <=4 mm^2) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain). Analysis after Vaccination 2 is only applicable for 6-35 months old group and 3-12 years old group.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33 | 33 | 33
percentage of participants
  A/H1N1: 21 days after Vaccination 1 (n=32,32,33) | 6.3 [0.766 to 20.807] | 81.3 [63.561 to 92.792] | 72.7 [54.476 to 86.700]
  A/H1N1: 21 days after Vaccination 2 (n=29,31,0) | 79.3 [60.275 to 92.006] | 90.3 [74.246 to 97.958] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  A/H3N2: 21 days after Vaccination 1 (n=32,32,33) | 18.8 [7.208 to 36.439] | 46.9 [29.094 to 65.256] | 42.4 [25.476 to 60.785]
  A/H3N2: 21 days after Vaccination 2 (n=29,31,0) | 69.0 [49.168 to 84.715] | 67.7 [48.627 to 83.318] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  B: 21 days after Vaccination 1 (n=32,32, 33) | 15.6 [5.275 to 32.788] | 62.5 [43.692 to 78.900] | 42.4 [25.476 to 60.785]
  B: 21 days after Vaccination 2 (n=29,31,0) | 48.3 [29.449 to 67.469] | 74.2 [55.387 to 88.144] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.

16. Secondary Outcome: GMFI in SRH Antibody Titer (Egg-Derived Antigen) From Baseline to 21 Days After Each Vaccination
Description: GMFI from baseline in SRH antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after each vaccination for all groups. Analysis after Vaccination 2 is only applicable for 6-35 months old group and 3-12 years old group.
Time Frame: Day 22 (21 days after Vaccination 1 for all groups), Day 43 (21 days after Vaccination 2 for 6 -35 months old group and 3-12 years old group)
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33 | 33 | 33
fold increase
  A/H1N1: 21 days after Vaccination 1 (n=32, 32, 33) | 1.2020 [0.98289 to 1.46989] | 2.4707 [1.89898 to 3.21447] | 2.7540 [1.97811 to 3.83430]
  A/H1N1: 21 days after Vaccination 2 (n=29, 31, 0) | 7.0652 [4.91411 to 10.15793] | 2.9292 [2.23349 to 3.84174] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  A/H3N2: 21 days after Vaccination 1 (n=32, 32, 33) | 1.5038 [1.18040 to 1.91588] | 1.9682 [1.57520 to 2.45935] | 2.0612 [1.51354 to 2.80709]
  A/H3N2: 21 days after Vaccination 2 (n=29, 31, 0) | 5.1163 [3.65073 to 7.17028] | 2.3363 [1.77098 to 3.08201] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  B: 21 days after Vaccination 1 (n=32, 32, 33) | 1.3443 [1.03252 to 1.75027] | 2.8400 [1.98458 to 4.06424] | 1.8889 [1.42420 to 2.50523]
  B:21 days after Vaccination 2 (n=29, 31, 0) | 3.7658 [2.66600 to 5.31917] | 3.8880 [2.72038 to 5.55686] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.

17. Secondary Outcome: GMT of SRH Antibody Titer (Egg-Derived Antigen)
Description: GMT of SRH antibody titer (egg-derived antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after each vaccination. Analysis after Vaccination 2 is only applicable for 6-35 months old group and 3-12 years old group.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33 | 33 | 33
titer
  A/H1N1: 21 days after Vaccination 1 (n=32, 32, 33) | 5.1604 [4.01580 to 6.63117] | 64.4700 [45.99985 to 90.35654] | 89.8328 [82.79308 to 97.47116]
  A/H1N1: 21 days after Vaccination 2 (n=29, 31, 0) | 30.5555 [21.50430 to 43.41647] | 83.8136 [74.30566 to 94.53822] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  A/H3N2: 21 days after Vaccination 1 (n=32, 32, 33) | 9.8918 [6.28974 to 15.55675] | 36.4508 [26.86516 to 49.45654] | 52.9301 [46.41297 to 60.36242]
  A/H3N2: 21 days after Vaccination 2 (n=29, 31, 0) | 33.0272 [24.40664 to 44.69260] | 46.7134 [37.50756 to 58.17885] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  B: 21 days after Vaccination 1 (n=32, 32, 33) | 6.3066 [4.34309 to 9.15778] | 41.4710 [29.47979 to 58.33961] | 70.2017 [58.66371 to 84.00902]
  B: 21 days after Vaccination 2 (n=29, 31, 0) | 16.9727 [11.66290 to 24.69991] | 52.8247 [44.14357 to 63.21315] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.

18. Secondary Outcome: Percentage of Participants With Seroprotection in HI Antibody Titer (Vero Antigen) of >=40
Description: Seroprotection rate was measured by HI antibody titer (Vero antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after each vaccination for all groups. Seroprotection rate was defined as the percentage of participants with HI antibody titer of >=40. Analysis after Vaccination 2 is only applicable for 6-35 months old group and 3-12 years old group.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33 | 33 | 33
percentage of participants
  A/H1N1: 21 days after Vaccination 1 (n=32, 32, 33) | 3.1 [0.079 to 16.217] | 90.6 [74.977 to 98.023] | 90.9 [75.668 to 98.085]
  A/H1N1: 21 days after Vaccination 2 (n=31, 31, 0) | 32.3 [16.682 to 51.373] | 93.5 [78.578 to 99.209] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  A/H3N2: 21 days after Vaccination 1 (n=32, 32, 33) | 28.1 [13.746 to 46.747] | 81.3 [63.561 to 92.792] | 97.0 [84.241 to 99.923]
  A/H3N2: 21 days after Vaccination 2 (n=31,31, 0) | 74.2 [55.387 to 88.144] | 87.1 [70.166 to 96.370] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  B: 21 days after Vaccination 1 (n=32, 32, 33) | 9.4 [1.977 to 25.023] | 34.4 [18.572 to 53.193] | 48.5 [30.796 to 66.456]
  B: 21 days after Vaccination 2 (n=31, 31, 0) | 9.7 [2.042 to 25.754] | 51.6 [33.061 to 69.845] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.

19. Secondary Outcome: Percentage of Participants With Seroconversion in HI Antibody Titer (Vero Antigen)
Description: Seroconversion rate was measured by HI antibody titer (Vero antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after each vaccination for all groups. Seroconversion rate was defined as the percentage of participants achieving a minimal 4-fold increase from baseline (with a baseline HI antibody titer of >=10), or achieving a HI antibody titer of >=40 (with baseline HI antibody titer of <10) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain). Analysis after Vaccination 2 is only applicable for 6-35 months old group and 3-12 years old group.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33 | 33 | 33
percentage of participants
  A/H1N1: 21 days after Vaccination 1 (n=32, 32, 33) | 0.0 [0.000 to 10.888] | 78.1 [60.027 to 90.723] | 69.7 [51.289 to 84.408]
  A/H1N1: 21 days after Vaccination 2 (n=31, 31, 0) | 32.3 [16.682 to 51.373] | 87.1 [70.166 to 96.370] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  A/H3N2: 21 days after Vaccination 1 (n=32, 32, 33) | 21.9 [9.277 to 39.973] | 43.8 [26.364 to 62.337] | 42.4 [25.476 to 60.785]
  A/H3N2: 21 days after Vaccination 2 (n=31,31, 0) | 67.7 [48.627 to 83.318] | 54.8 [36.034 to 72.684] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  B: 21 days after Vaccination 1 (n=32, 32, 33) | 9.4 [1.977 to 25.023] | 28.1 [13.746 to 46.747] | 42.4 [25.476 to 60.785]
  B: 21 days after Vaccination 2 (n=31, 31, 0) | 9.7 [2.042 to 25.754] | 48.4 [30.155 to 66.939] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.

20. Secondary Outcome: GMFI in HI Antibody Titer (Vero Antigen) From Baseline to 21 Days After Each Vaccination
Description: GMFI from baseline in HI antibody titer (Vero antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after each vaccination for all groups. Analysis after Vaccination 2 is only applicable for 6-35 months old group and 3-12 years old group.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33 | 33 | 33
fold increase
  A/H1N1: 21 days after Vaccination 1 (n=32, 32, 33) | 1.02 [0.978 to 1.068] | 16.17 [9.606 to 27.233] | 7.51 [4.800 to 11.754]
  A/H1N1: 21 days after Vaccination 2 (n=31, 31, 0) | 2.30 [1.472 to 3.592] | 17.30 [10.589 to 28.268] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  A/H3N2: 21 days after Vaccination 1 (n=32, 32, 33) | 1.72 [1.264 to 2.338] | 3.67 [2.250 to 5.979] | 3.90 [2.387 to 6.361]
  A/H3N2: 21 days after Vaccination 2 (n=31, 31, 0) | 6.40 [4.110 to 9.954] | 4.78 [2.937 to 7.791] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  B: 21 days after Vaccination 1 (n=32, 32, 33) | 1.27 [0.965 to 1.669] | 2.62 [1.695 to 4.055] | 3.21 [2.130 to 4.833]
  B: 21 days after Vaccination 2 (n=31, 31, 0) | 1.28 [0.964 to 1.697] | 2.99 [1.918 to 4.663] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.

21. Secondary Outcome: GMT of HI Antibody Titer (Vero Antigen)
Description: GMT of HI antibody titer (Vero antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after each vaccination. Analysis after Vaccination 2 is only applicable for 6-35 months old group and 3-12 years old group.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33 | 33 | 33
titer
  A/H1N1: 21 days after Vaccination 1 (n=32, 32, 33) | 5.34 [4.673 to 6.092] | 156.57 [99.959 to 245.257] | 69.79 [49.992 to 97.430]
  A/H1N1: 21 days after Vaccination 2 (n=31, 31, 0) | 12.03 [7.571 to 19.101] | 187.11 [123.079 to 284.443] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  A/H3N2: 21 days after Vaccination 1 (n=32, 32, 33) | 16.46 [8.314 to 32.578] | 94.11 [50.943 to 173.861] | 141.80 [102.494 to 196.169]
  A/H3N2: 21 days after Vaccination 2 (n=31, 31, 0) | 62.55 [34.861 to 112.233] | 143.08 [79.875 to 256.286] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  B: 21 days after Vaccination 1 (n=32, 32, 33) | 6.35 [4.825 to 8.344] | 15.26 [9.688 to 24.026] | 19.38 [12.917 to 29.076]
  B: 21 days after Vaccination 2 (n=31, 31, 0) | 6.39 [4.819 to 8.483] | 17.49 [10.923 to 28.003] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.

22. Secondary Outcome: Percentage of Participants With Seroprotection in SRH Antibody Titer (Vero Antigen) of >= 25 mm^2
Description: Seroprotection rate was measured by SRH antibody titer (Vero Antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after each vaccination for all groups. Seroprotection rate was defined as the percentage of participants with SRH antibody titer of >=25 mm^2. Analysis after Vaccination 2 is only applicable for 6-35 months old group and 3-12 years old group.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33 | 33 | 33
percentage of participants
  A/H1N1: 21 days after Vaccination 1 (n=32, 32, 33) | 0.0 [0.000 to 10.888] | 75.0 [56.595 to 88.538] | 81.8 [64.540 to 93.021]
  A/H1N1: 21 days after Vaccination 2 (n=29, 31, 0) | 10.3 [2.186 to 27.352] | 87.1 [70.166 to 96.370] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  A/H3N2: 21 days after Vaccination 1 (n=32, 32, 33) | 34.4 [18.572 to 53.193] | 90.6 [74.977 to 98.023] | 97.0 [84.241 to 99.923]
  A/H3N2: 21 days after Vaccination 2 (n=29, 31, 0) | 86.2 [68.336 to 96.111] | 96.8 [83.298 to 99.918] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  B: 21 days after Vaccination 1 (n=32, 32, 33) | 15.6 [5.275 to 32.788] | 71.9 [53.253 to 86.254] | 81.8 [64.540 to 93.021]
  B: 21 days after Vaccination 2 (n=29, 31, 0) | 27.6 [12.734 to 47.238] | 83.9 [66.273 to 94.548] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.

23. Secondary Outcome: Percentage of Participants With Seroconversion in SRH Antibody Titer (Vero Antigen)
Description: Seroconversion rate was measured by SRH antibody titer (Vero antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after each vaccination for all groups. Seroconversion rate was defined as the percentage of participants achieving a minimal 50% increase from baseline (with a baseline SRH antibody titer of >4 mm^2), or achieving a SRH antibody titer of >=25 mm^2 (with baseline SRH antibody titer of <=4 mm^2) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain). Analysis after Vaccination 2 is only applicable for 6-35 months old group and 3-12 years old group.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33 | 33 | 33
percentage of participants
  A/H1N1: 21 days after Vaccination 1 (n=32, 32, 33) | 0.0 [0.000 to 10.888] | 75.0 [56.595 to 88.538] | 54.5 [36.351 to 71.893]
  A/H1N1: 21 days after Vaccination 2 (n=29, 31, 0) | 10.3 [2.186 to 27.352] | 87.1 [70.166 to 96.370] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  A/H3N2: 21 days after Vaccination 1 (n=32, 32, 33) | 18.8 [7.208 to 36.439] | 40.6 [23.698 to 59.355] | 51.5 [33.544 to 69.204]
  A/H3N2: 21 days after Vaccination 2 (n=29, 31, 0) | 72.4 [52.762 to 87.266] | 58.1 [39.076 to 75.452] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  B: 21 days after Vaccination 1 (n=32, 32, 33) | 12.5 [3.513 to 28.995] | 56.3 [37.663 to 73.636] | 57.6 [39.215 to 74.524]
  B: 21 days after Vaccination 2 (n=29, 31, 0) | 24.1 [10.298 to 43.540] | 64.5 [45.370 to 80.773] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.

24. Secondary Outcome: GMFI in SRH Antibody Titer (Vero Antigen) From Baseline to 21 Days After Each Vaccination
Description: GMFI from baseline in SRH antibody titer (Vero antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after each vaccination for all groups. Analysis after Vaccination 2 is only applicable for 6-35 months old group and 3-12 years old group.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33 | 33 | 33
fold increase
  A/H1N1: 21 days after Vaccination 1 (n=32, 32, 33) | 1.0000 [NA to NA] — 95% confidence interval was not calculable because SRH antibody titers of Pre-vaccination and Post-vaccinations in all participants were same. | 3.8815 [2.91105 to 5.17543] | 3.0063 [2.06690 to 4.37270]
  A/H1N1: 21 days after Vaccination 2 (n=29, 31, 0) | 1.2706 [0.99257 to 1.62639] | 4.1427 [3.11949 to 5.50159] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  A/H3N2: 21 days after Vaccination 1 (n=32, 32, 33) | 1.4480 [1.18483 to 1.76972] | 1.7522 [1.41051 to 2.17678] | 2.0947 [1.57731 to 2.78168]
  A/H3N2: 21 days after Vaccination 2 (n=29, 31, 0) | 4.9597 [3.52649 to 6.97548] | 2.2506 [1.67926 to 3.01629] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  B: 21 days after Vaccination 1 (n= 32, 32, 33) | 1.2209 [0.97777 to 1.52445] | 3.6157 [2.38627 to 5.47866] | 2.6846 [1.92487 to 3.74409]
  B:21 days after Vaccination 2 (n= 29, 31, 0) | 2.2979 [1.59954 to 3.30117] | 4.4759 [3.05031 to 6.56777] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.

25. Secondary Outcome: GMT of SRH Antibody Titer (Vero Antigen)
Description: GMT of SRH antibody titer (Vero antigen) for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after each vaccination. Analysis after Vaccination 2 is only applicable for 6-35 months old group and 3-12 years old group.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Number analyzed (Participants) | 33 | 33 | 33
titer
  A/H1N1: 21 days after Vaccination 1 (n=32, 32, 33) | 4.0000 [NA to NA] — 95% confidence interval was not calculable because SRH antibody titers of Pre-vaccination and Post-vaccinations in all participants were same. | 26.8737 [20.52041 to 35.19414] | 32.3664 [25.74333 to 40.69349]
  A/H1N1: 21 days after Vaccination 2 (n=29, 31, 0) | 5.0822 [3.97027 to 6.50558] | 30.9216 [24.14566 to 39.59911] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  A/H3N2: 21 days after Vaccination 1 (n=32, 32, 33) | 12.2879 [8.09586 to 18.65065] | 40.3869 [31.13697 to 52.38484] | 61.7091 [53.35048 to 71.37721]
  A/H3N2: 21 days after Vaccination 2 (n=29, 31, 0) | 40.4564 [32.19850 to 50.83224] | 55.3238 [48.82904 to 62.68238] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.
  B: 21 days after Vaccination 1 (n=32, 32, 33) | 6.5038 [4.44742 to 9.51111] | 35.8443 [25.16079 to 51.06422] | 38.2075 [29.71344 to 49.12974]
  B: 21 days after Vaccination 2 (n=29, 31, 0) | 10.8420 [7.20922 to 16.30540] | 44.8583 [36.23158 to 55.53899] | NA [NA to NA] — Data is not required for this age group because Vaccination 2 is not planned for 13-19 years old group.

ADVERSE EVENTS:
Time Frame: TAEs are AEs, regardless of relationship to drug, that occur or worsen after first dose of study vaccine and no more than 21 days after the last dose (up to Day 43 for 6-35 months old group and 3-12 years old group, up to Day 22 for 13-19 years old group)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-850 0.25 mL: 6-35 Months | TAK-850 0.5 mL: 3-12 Years | TAK-850 0.5 mL: 13-19 Years
Serious Adverse Events (participants affected / at risk) | 0/33 | 1/33 | 0/33
Other Adverse Events (participants affected / at risk) | 21/33 | 29/33 | 24/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-850 0.25 mL: 6-35 Months (N=33) | TAK-850 0.5 mL: 3-12 Years (N=33) | TAK-850 0.5 mL: 13-19 Years (N=33)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-850 0.25 mL: 6-35 Months (N=33) | TAK-850 0.5 mL: 3-12 Years (N=33) | TAK-850 0.5 mL: 13-19 Years (N=33)
Eye discharge (Eye disorders) | 4 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 2
Injection site pain (General disorders) | 3 | 24 | 19
Pyrexia (General disorders) | 12 | 3 | 1
Injection site swelling (General disorders) | 0 | 6 | 3
Malaise (General disorders) | 0 | 5 | 3
Injection site erythema (General disorders) | 0 | 6 | 1
Fatigue (General disorders) | 0 | 4 | 2
Injection site haemorrhage (General disorders) | 4 | 1 | 0
Injection site induration (General disorders) | 0 | 3 | 2
Injection site pruritus (General disorders) | 0 | 4 | 1
Injection site warmth (General disorders) | 0 | 4 | 0
Crying (General disorders) | 2 | 1 | 0
Irritability postvaccinal (General disorders) | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 3
Molluscum contagiosum (Infections and infestations) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Somnolence (Nervous system disorders) | 5 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi-site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.